CLINICAL TRIAL: NCT01614093
Title: Effects of Intranasal Oxytocin on Satiety Signaling in People With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, Dr. Kimberly Warren, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00049602
Record Dates: First submitted 2012-03-20; First posted 2012-06-07 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Appetite; Oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: All participants will receive both active drug and placebo, differences between treatment conditions will be analyzed due to small sample order effects will not be analyzed
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin/Placebo (Active Comparator): Each participant will receive intranasal oxytocin 24IU or intranasal saline 24IU in random order. All results will be reported by treatment, the sample is too small for order effects.
  Interventions: Drug: Oxytocin; Drug: Placebo
- Placebo/Oxytocin (Active Comparator): Each participant will receive intranasal oxytocin 24IU or intranasal saline 24IU in random order. All results will be reported by treatment, the sample is too small for order effects.
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Single dose intranasal oxytocin (24 IU)
Drug: Placebo — Placebo- Sugar pill

SUMMARY:
The objective of this study is to test a single dose of intranasal oxytocin, compared to placebo, in a within subjects, crossover design, to see if oxytocin will improve satiety signaling (behaviorally and/or by self report) compared to placebo. If this single dose pilot paradigm shows an increase in satiety, it may be tested in follow-up studies as a prevention or treatment for weight gain and overeating in people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Male or Female
* Age: 18 to 54 years
* Caucasian or Non-Caucasian
* Body Mass Index of ≥ 27 kg/m2
* One month of stable antipsychotic treatment (same medication regimen and same dose)

Exclusion Criteria:

* History of organic brain disease
* DSM-IV diagnosis of Mental Retardation
* DSM-IV diagnosis of Alcohol or Substance Dependence within the last six months (except nicotine)
* DSM-IV diagnosis of Alcohol or Substance Abuse within the last one month (except nicotine)
* Are pregnant or lactating
* Meet DSM-IV criteria for a past and/or current eating disorder via the SCID, or if they have a past medical history of an eating disorder, received treatment/counseling for an eating disorder and/or required hospitalization for an eating disorder. (If an otherwise undiagnosed eating disorder is detected during screening, referral to treatment will be provided.)
* Are taking weight-loss medications, whether over-the-counter (i.e. Hydroxycut, Stacker products, Metabo-Plus, CortiSlim), or prescribed, including appetite suppressants (Didrex, Tenuate, Sanorex, Mazanor, Adipex-P, Meridia, and Phentermine) and fat-absorption inhibitors (Xenical).
* Have cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires. This is defined an as a score of less than 10 on the Evaluation to Sign Consent (ESC).
* Have a medical illness, dietary restrictions, or food allergies that, in the view of the investigators, would compromise participation.
* Are taking prostaglandins such as dinoprostone or misoprostol (because they interact with oxytocin).

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Warren, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- See also: Related Info — http://www.mprc.umaryland.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants were randomized, 16 participants participated in the trial. All data is available for only 16 participants
Groups:
- Oxytocin/ Placebo: Each participant will receive intranasal oxytocin 24IU or intranasal saline 24IU in random order. All results will be reported by treatment, the sample is too small for order effects.
Period: Overall Study
Arm/Group | Oxytocin/ Placebo
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Oxytocin vs Placebo: Participants rated themselves as significantly less hungry when administered OT (M=36.37, SD=21.0) than placebo (M=44.81, SD=28.6) at 60 min. post-preload, F(5, 15)=8.05, p=0.012.
Arm/Group | Oxytocin vs Placebo
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 32 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 7
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Food Consumption After Intervention
Description: We hypothesize that participants will have greater satiety signaling, indicated by less consumption of the "Test Meal" consumed 90 minutes after the preload.
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: Grams
Groups:
- Oxytocin/Placebo: Each participant received intranasal oxytocin 24IU or intranasal saline 24IU in random order. All results will be reported by treatment, the sample is too small for order effects.
Arm/Group | Oxytocin/Placebo
Number analyzed (Participants) | 16
Grams
  Oxytocin | 7.9 (13.0)
  Placebo | 7.4 (12.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of about 4 weeks (on each of the visit days)
Groups:
- Oxytocin; Placebo: Each participant will receive intranasal oxytocin 24IU or intranasal saline 24IU in random order. All results will be reported by treatment, the sample is too small for order effects.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxytocin (N=16) | Placebo (N=16)
Loss of Appetite (General disorders) | 1 | 1
Bruisng Easily (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dizziness (General disorders) | 1 | 0
Enuresis (General disorders) | 0 | 1
Malise (General disorders) | 0 | 1
Hyersalavation (General disorders) | 0 | 1
Sedation (General disorders) | 1 | 2
Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No